CLINICAL TRIAL: NCT06522243
Title: Effectiveness of Mindfulness Program for Parents of Children With SEN
Brief Title: Mindful Parenting for Parents With SEN Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, XU Jia-Qi Melody, Senior Professional Practitioner, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA240327
Record Dates: First submitted 2024-07-15; First posted 2024-07-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Expressed Emotion; Stress; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: waitlist randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- immediate intervention (Experimental): Start with the 8-week intervention immediately/soon after recruitment
  Interventions: Behavioral: 8-week mindful parenting program
- waitlist control (No Intervention): No intervention while being assessed but will receive the intervention after the assessments

INTERVENTIONS:
Behavioral: 8-week mindful parenting program — The current study adopts the Mindful Parenting program developed by Prof Susan Bögels (Bögels & Restifo, 2013), which is an application of mindfulness-based intervention which aims to improve parenting by reducing parents' own stress levels, decreasing parental automatic reactivity, increasing open and unbiased attitudes towards children, and decreasing inter-generational dysfunctional parenting (Bögels et al., 2014). The program consists of eight consecutive weeks of parent groups and one follow-up session two months after the last session. Each parent group will include 15-20 participants. The original Mindful Parenting Program will last for around 3 hours for each session, with the longest practice of 40 minutes. Considering parents recruited in the study may have a higher risk of psychiatric conditions than the general population, each session of mindful parenting group will be reduced to 2 to 2.5 hours with the longest mindfulness practice of 30 minutes (Baer et al., 2019).
  Arms: immediate intervention

SUMMARY:
The goal of the study is to evaluate the effectiveness of an online eight-week mindful parenting program for parents of adolescents with special needs and its impact on parents' wellbeing and behaviors of their adolescents with SEN(s).

Researchers will randomize the participants into the immediate intervention group (to start the intervention soon after recruitment) and the waitlist control group (to start the intervention after the immediate intervention group) so as to compare the changes between the two groups.

The participants will join the 8-week mindful parenting intervention and one follow-up session. They will be asked to fill in the questionnaires at baseline, after the 8-week intervention, and at the follow-up sessions. Training sessions will be audio-taped and transcripted. The conversation during the zoom classes and participants' sharing on their subjective experience related to mindfulness practices will be analysed.

DETAILED DESCRIPTION:
Being a parent is inherently a demanding and stressful job, and raising children with SEN may pose additional stressors to parents. Parents of SEN children have higher parenting stress compared to those of typically developed children in facing daily challenges with their children's learning and development, which may lead to a higher risk of child maltreatment. Adolescence and emerging adulthood are a transition period which may impose increased stress and challenges on both young people and their parents. As a result, parents of young people with SEN(s) require more support in both parenting skills and their own psychological wellbeing.

Parents not only provide care for their children but also create an everyday environment under which their children are raised. Improvements in parenting skills and parents' mental health could lead to positive outcomes for child and youth mental wellbeing (while malfunctioning parenting may also impose an aversive effect on children's development. For instance, a critical and over-involvement of parental-child interaction, i.e., high expressed emotion (high EE) in the family, was found to be a robust predictor of relapse in different psychiatric illnesses.

Parenting is by nature a highly challenging and complex job and raising a child with mental illness could be even more stressful and strain parents' experience. It was reported that the severity of children's emotional and behavioral disturbances was closely related to parents' stress levels. On the other hand, parenting stress is an essential factor contributing to parenting effectiveness. When parents experience a high level of stress, their parenting effectiveness may decrease. Hence, reducing parents' stress levels would not only benefit parents themselves but also enhance effective parenting so as to benefit the wellbeing of their children with mental illness.

Mindful parenting Mindful parenting has been defined as the ability to pay attention to your children and parenting in an intentional, non-judgmental, and moment-to-moment awareness. Mindful parenting intervention does not directly teach parenting skills like other parenting training programs. Being mindful in everyday parenting is to perceive their children with an unbiased and open attitude, providing more sensible and responsive reactions to the children instead of reacting automatically based on past experience of parenting or being parented. By decentering from the current thoughts or affects, it enables parents to observe their internal experiences objectively without overidentifying with them. This, in turn, strengthens their capacity to endure the intense emotions and allow them to be more fully present with their child. Mindful parenting was also found to be negatively correlated with parental stress, yet positively associated with the levels of adopting authoritative parenting style. Furthermore, one of the features of the mindful parenting program is to practice non-judgmental awareness when interacting with children instead of automatically reacting to children's behaviours. It is thus speculated that mindful parenting practice could also promote less high EE interactions between parents and adolescents, which has been sparsely studied in the existing literature. The current pilot study may thus provide a possible mechanism in explaining the effectiveness of mindful parenting in improving the wellbeing of both parents and their children with SEN(s).

Mindful parenting had been applied in parenting for children with special needs, childbirth and parenting, and parenting for children with mental illness. The results of various mindful parenting programs (with a minimum of 6-8 weekly group sessions) showed some evidence of improvements for parenting stress, parents' psychopathology, and their children's mental health symptoms. However, the study sample had mainly focused on parents whose children were in their early or middle childhood.

The current study thus aims to recruit a more diverse sample of adolescents with different types of SENs. The data and experience gained from the current pilot study would also shed light on a clearer picture of whether a nine-session mindful parenting program would benefit both parents and their adolescent children with SENs.

A mixed methods design with qualitative journaling and quantitative experimental design could leverage the benefits of both methods. The data collected from participants' journal writing would elucidate the benefits, challenges, and personal growth through mindfulness practices from a subjective experiential perspective. It will also provide valuable insights for designing a larger-scale study to understand the underlying mechanism of mindful parenting on wellbeing of both parents and their children with SEN.

Aims and Hypotheses to be Tested:

The current study aims to (i) to evaluate the effectiveness of mindfulness training in enhancing the wellbeing of both parents and behaviors of their adolescents with SEN(s); (ii) to assess the feasibility and acceptability of adopting a nine-session Mindful Parenting program among parents of adolescents with SEN(s); (iii) to formulate useful suggestions and guidelines on mindfulness training for parents of adolescents with SEN(s).

ELIGIBILITY:
Inclusion Criteria:

* with one adolescent child with special educational need(s)
* being the major caregiver for the adolescent for at least one year
* Cantonese speaker

Exclusion Criteria:

* schizophrenia-spectrum disorder
* bipolar disorder
* substance abuse
* developmental disabilities
* physical disabilities
* with active psychotic symptoms
* high suicidal risks
* experiencing a recent personal crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Parental Stress | 16 weeks
  Parental Stress Scale is an 18-item self-report measure in which parents respond to statements about their typical relationship with their child. For each statement, respondents rate their level of agreement on a 5-point Likert scale (1- strongly disagree, 2 - disagree, 3- undecided, 4 - agree, and 5 -strongly agree).Higher scores reflect more parental stress. The possible range of the PSS is 18 (low stress) to 90 (high stress).
Mindfulness in Parenting | 16 weeks
  The 31-item Chinese version of the Interpersonal Mindfulness in Parenting Scale (IM-P) will be used to evaluate parents' mindfulness on four aspects, including compassion for the child, nonjudgmental acceptance in parenting, emotional awareness, and listening with full attention. A total sum will be calculated to indicate mindfulness in parenting with a higher score implying better outcome (minimum value=31; maximum value=155).
Parents' Expressed Emotion | 16 weeks
  Family Questionnaire (FQ) is used to evaluate the parents' level of expressed emotion, including criticism and over-involvement. FQ is a 20-item parent self-rated questionnaire with four possible answers ranging from "never/very rarely" to "very often." A total score will be calculated with a higher score indicating a a higher level of expressed emotion (minimum value=20; maximum value=80).
Children's behaviors | 16 weeks
  The 25-item Chinese version of the Strength and Difficulties Questionnaire (SDQ) will be used to assess the externalising and internalising problems of adolescents. It comprises five subscales, ranging from emotional problems, conduct problems, hyperactivity, peer problems and prosocial behaviours in adolescents. Each item is rated on a Likert scale from 0 (not true) to 2 (certainly true). A total difficulties score will be calculated with a higher score implying more difficult behaviors by summing scores from all the items except the prosocial scale (minimum value=0; maximum value=40).

SECONDARY OUTCOMES:
General Mindfulness Awareness | 16 weeks
  To assess the general mindfulness awareness in parents, the short 15-item version of the Five Facet Mindfulness Questionnaire (FFMQ-15) will be used. A total sum will be calculated to indicate trait mindfulness with a higher score implying better outcome (minimum value=15; maximum value=75).
Decentering | 16 weeks
  Decentering is measured using the Experiences Questionnaire, an 11-item self-report scale that assesses the construct of decentering or disidentification with content of negative thinking. A total sum will be calculated to indicate level of decentering with a higher score implying better outcome (minimum value=5; maximum value=55).
Parenting Skills | 16 weeks
  Alabama Parenting Questionnaire-short version is a 9-item self-rated questionnaire used to measures three factors in parenting: positive parenting, inconsistent discipline and poor supervision. Items are scored from 1 (never) to 5 (always). A higher score in subscale of positive parenting (minimum value=3; maximum value=15) indicates a better outcome while a higher score in subscales of inconsistent discipline and poor supervision (minimum value=3; maximum value=15) indicate worse outcomes.

OTHER OUTCOMES:
Subjective experiences with mindful parenting | 16 weeks
  Training sessions will be audio-taped and transcripted. The conversation during the zoom classes and participants' sharing on their subjective experience related to mindfulness practices will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Xu Jia-QI, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kogure H. [Brain metabolism disorder associated with cerebral ischemia]. Nihon Rinsho. 1985 Feb;43(2):349-60. No abstract available. Japanese. PMID 2987569
- [Background] Shiba R, Sakoda S, Yamada N. Peripheral ameloblastoma. J Oral Maxillofac Surg. 1983 Jul;41(7):460-3. doi: 10.1016/0278-2391(83)90132-5. PMID 6575147
- [Background] Butzlaff RL, Hooley JM. Expressed emotion and psychiatric relapse: a meta-analysis. Arch Gen Psychiatry. 1998 Jun;55(6):547-52. doi: 10.1001/archpsyc.55.6.547. PMID 9633674
- [Background] Crijnen AA, Achenbach TM, Verhulst FC. Problems reported by parents of children in multiple cultures: the Child Behavior Checklist syndrome constructs. Am J Psychiatry. 1999 Apr;156(4):569-74. doi: 10.1176/ajp.156.4.569. PMID 10200736
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] van der Oord S, Bogels SM, Peijnenburg D. The Effectiveness of Mindfulness Training for Children with ADHD and Mindful Parenting for their Parents. J Child Fam Stud. 2012 Feb;21(1):139-147. doi: 10.1007/s10826-011-9457-0. Epub 2011 Feb 2. PMID 22347788
- [Background] Wiedemann G, Rayki O, Feinstein E, Hahlweg K. The Family Questionnaire: development and validation of a new self-report scale for assessing expressed emotion. Psychiatry Res. 2002 Apr 15;109(3):265-79. doi: 10.1016/s0165-1781(02)00023-9. PMID 11959363
- [Background] Xu JQ, Poon K, Ho MSH. Brief Report: The Impact of COVID-19 on Parental Stress and Learning Challenges for Chinese Children with SpLD. J Autism Dev Disord. 2025 Jun;55(6):2186-2193. doi: 10.1007/s10803-023-05983-y. Epub 2023 Apr 20. PMID 37079179